CLINICAL TRIAL: NCT05027165
Title: Prospective Evaluation of Immunological, Molecular-genetic, Image-based and Microbial Analyzes to Characterize Tumor Response and Control in Patients With Inoperable Stage III NSCLC Treated With Chemoradiotherapy Followed by Consolidation Therapy With Durvalumab (PRECISION)
Brief Title: Prospective Evaluation of Immunological, Molecular-genetic, Image-based and Microbial Analyzes to Characterize Tumor Response and Control in Patients With Inoperable Stage III NSCLC Treated With Chemoradiotherapy Followed by Consolidation Therapy With Durvalumab
Acronym: PRECISION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: LMU Klinikum (Other)
Collaborators: Department of Internal Medicine V, Thoracic Oncology Centre Munich, LMU Munich, Munich, Germany (Unknown); Institute of Pathology, Faculty of Medicine, LMU Munich, Munich, Germany (Unknown); Asklepios Lung Clinic, Munich-Gauting, Germany (Unknown); Department of Radiology, University Hospital, LMU Munich, Munich, Germany (Unknown); Department of Nuclear Medicine, University Hospital, LMU Munich, Munich, Germany (Unknown); Institute for Medical Information Processing, Biometry and Epidemiology, LMU München, Munich, Germany (Unknown); Department of Medicine II, University Hospital, LMU Munich, Munich, Germany (Unknown); Immunoanalytics Research Group Tissue Control of Immunocytes, Helmholtz Center Munich, Munich, Germany (Unknown)
Responsible Party: Principal Investigator, Farkhad Manapov, PD Dr. med Farkhad Manapov, LMU Klinikum
Other Study IDs: 20-502
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Oncology; Biomarker; NSCLC, Stage III; Durvalumab; Chemoradiotherapy
Keywords: NSCLC; Stage III; Biomarker
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Short circulating tumor total nucleic acid (ctTNA: ctDNA and ctRNA) within blood sample and possible mutations will be analysed at six different time points (blood sample will be collected 5-10 d before, after 15 fractions, at the end of concurrent chemoradiotherapy as well as 3-, 6- and 12 months after start of durvalumab).
  Blood samples will be evaluated using the Oncomine Pan-Cancer Cell free Assay (Life Technololgies) NGS (next generation sequencing).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: In this cohort, 40 NSCLC patients with indication for chemoradiotherapy followed by durvalumab maintenance treatment ("standard of care") will be consecutively recruited.
  Comprehensive characterization of all patients includes immunophenotyping of peripheral blood mono-nuclear cells, ctDNA as well as gut/saliva microbiome analyses and will be performed before, after 15 fractions of radiotherapy, at the end of concurrent chemoradiotherapy as well as 3-, 6- and 12 months after start of durvalumab.
  18F-FDG-PET/CT will be performed 5-10 d before start of radiotherapy, 6 weeks, 6 months,12 and 24 months after the end of radiochemotherapy. Lung function will be asssed before start of radiotherapy, at the end and 6 weeks after chemoradiotherapy as well as 3-, 6- and 12, 18, 24months after start of durvalumab.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — No intervention

SUMMARY:
This non-interventional single-center explorative biomarker study aims at longitudinal comprehensive characterization (molecular genetics, immunological, morphological, image-based and microbial features) of the patient (host) and tumor as well as changes during standard treatment and in case of recurrent disease in inoperable stage III non-small cell lung cancer (NSCLC). Comprehensive analysis will include peripheral blood cellular and humoral immunophenotyping, circulating tumor DNA and gut/saliva microbiota analyses. 18F-FDG-PET/CT before, 6 weeks, 6- and 12-months after chemoradiotherapy as well as daily in course of radiation treatment cone-beam-CT and/or MRI imaging are included for morphological analysis. This study will provide valuable information of predictive biomarkers in patients with stage III NSCLC treated with durvalumab maintenance treatment after concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
The study will enrol 40 patients with stage III inoperable non-small cell lung cancer (NSCLC) who received standard chemoradiotherapy followed by maintenance therapy with PD-L1 inhibition (durvalumab) according to the current European Medicines Agency (EMA) approval.

The oncological treatment is carried out according to the international standards of radiation oncology/medical oncology. These are implemented by the department of radiation oncology at the University Hospital Munich (LMU) in their SOPs. Therefore, all patients will be treated with concurrent platinum-based chemoradiotherapy followed by durvalumab maintenance treatment 12 months after the end of chemoradiotherapy at the department of radiation oncology (University Hospital Munich (LMU)). Comprehensive characterization of all patients includes immunophenotyping of peripheral blood mono-nuclear cells, ctDNA as well as gut/saliva microbiome analyses and will be performed before, after 15 fractions of radiotherapy, at the end of concurrent chemoradiotherapy as well as 3-, 6- and 12 months after start of durvalumab.

18F-FDG-PET/CT will be performed 5-10 d before start of radiotherapy, 6 weeks, 6 months,12 and 24 months after the end of chemoradiotherapy. Lung function will be assessed before start of radiotherapy, at the end and 6 weeks after chemoradiotherapy as well as 3-, 6- and 12, 18, 24 months after start of durvalumab.

Follow-up will be performed by the department of radiation oncology at the University Hospital Munich (LMU) according to the clinical SOPs.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Histologically/cytologically confirmed diagnosis of non-small-cell lung cancer (NSCLC)
* Patients with non-operable NSCLC in tumor stage III A/B/C after UICC 8
* Eligible for platinum-based concurrent chemoradiotherapy followed by durvalumab maintenance treatment
* No invasive carcinoma in the last five years.
* ECOG Performance Status 0-2
* Lung function parameters (before or after bronchodilation): FEV1 ≥ 1.0 L and/or DLCO-SB ≥ 40%
* A maximum of two cycles of induction chemotherapy are permissible before start of chemoradiotherapy

Exclusion Criteria:

* Simultaneous participation in another clinical trial
* Mixed histology of small-cell and non-small-cell lung cancer
* Brain metastases confirmed by a contrast enhanced cMRI
* Prior receipt of an immunotherapy or investigational medicinal product
* Previous exposure to an anti-PD-1 or anti-PD-L1 antibody
* Pneumonitis ≥ Grade 2 as a result of prior radio-/chemoradiotherapy
* Patients with a non-active disease in the last 5 years can be included, but only after consultation with the responsible investigator of the study or his representative
* Primary immunodeficiencies in previous history
* Prior Interstitial lung disease (ILD)
* Prior autoimmune disease
* Previous organ transplantation with subsequent therapeutic immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enrol 40 patients with stage III inoperable non-small cell lung cancer (NSCLC) who received standard chemoradiotherapy followed by maintenance therapy with PD-L1 inhibition (durvalumab) at the department of radiation oncology, University Hospital Munich (LMU).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-11-07 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Predictive biomarker for progression-free survival at 12 and 24 months | 24 months
  To identify early immunological and morphological biomarkers and their dynamic changes to predict progression-free survival at 12 and 24 months.

SECONDARY OUTCOMES:
Predictive biomarkers for progression-free survival, overall survival, response rate, local and distant tumor control | 24 months
  To identify predictive biomarkers for progression-free survival at 6 and 18 months after chemoradiotherapy and overall survival and response rate, local and distant tumor control at 6 weeks, 6-, 12-, 18 and 24 months from the end of chemoradiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Farkhad Manapov, PhD MD, Principal Investigator — LMU University hospital, Munich, Germany
Locations (1):
- LMU University Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Data is available on request due to privacy/ethical restrictions.

REFERENCES:
- [Derived] Kasmann L, Taugner J, Eze C, Nieto A, Pelikan C, Florsch B, Kenndoff S, Hofer TP, Nossner E, Schulz C, Unterrainer M, Tufman A, Klauschen F, Jung A, Neumann J, Kumbrink J, Reinmuth N, Bartenstein P, Belka C, Manapov F. Prospective evaluation of immunological, molecular-genetic, image-based and microbial analyses to characterize tumor response and control in patients with unresectable stage III NSCLC treated with concurrent chemoradiotherapy followed by consolidation therapy with durvalumab (PRECISION): protocol for a prospective longitudinal biomarker study. Transl Lung Cancer Res. 2022 Jul;11(7):1503-1509. doi: 10.21037/tlcr-21-1010. PMID 35958344